CLINICAL TRIAL: NCT02403804
Title: Dietary Supplementation to Increase Serum Choline Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-1783; UL1TR001082 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-03-31 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Dietary supplements; serum choline; women
MeSH Terms: interventions — Phosphatidylcholines; Betaine; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Other): All 3 weeks will occur during luteal phase of menstrual cycle with a two-to-three week washout period between weeks.
  Week 1: Phosphatidylcholine 3600 mg qam and 2700 mg qpm
  Week 2: Betaine anhydrous 588 mg qam and 412 mg qpm
  Week 3: Betaine anhydrous 1000 mg BID
  Interventions: Dietary Supplement: Phosphatidylcholine; Dietary Supplement: Betaine (588 mg qam and 412 mg qpm); Dietary Supplement: Betaine (1000 mg BID)

INTERVENTIONS:
Dietary Supplement: Phosphatidylcholine — Phosphatidylcholine 3600 mg qam and 2700 mg qpm
Dietary Supplement: Betaine (588 mg qam and 412 mg qpm) — Betaine anhydrous 588 mg qam and 412 mg qpm
  Other Names: Trimethylglycine
Dietary Supplement: Betaine (1000 mg BID) — Betaine anhydrous 1000 mg BID
  Other Names: Trimethylglycine

SUMMARY:
The goal is to assess whether, in adult women during the luteal phase of their menstrual cycle, supplementing their diet with either phosphatidylcholine or betaine increases their serum choline levels.

DETAILED DESCRIPTION:
Elevated maternal serum free choline has the potential to improve fetal brain development . However, in humans, choline can be metabolized by gut flora into two metabolites with adverse outcomes: trimethylurea (which causes body odor) and Trimethylamine (TMA) which is then, once absorbed, metabolized into Trimethylamine-N-Oxide (TMAO). There is some concern that TMAO may be atherogenic and thus, if elevated over an extended period of time, may increase risk for cardiac disease. Thus, while maternal choline supplementation may improve fetal brain development, there is a potential for maternal adverse effects.

However, humans have an active choline metabolic pathway, and other components of the choline metabolic pathway (e.g. phosphatidylcholine and betaine) may be interchangeable with choline post absorption but are resistant to gut bacteria metabolism (i.e. serum TMA does not increase). Thus, these other compounds would be expected to increase serum but with no impact on TMA or trimethylurea levels. An initial study of phosphatidylcholine supplementation in pregnant women was consistent with this hypothesis; infant offspring demonstrated improved cerebral inhibition; while no adverse events were identified for either mother or infant.

Unfortunately, because of the lipid groups incorporated into phosphatidylcholine, its molecular weight is high and reasonable doses require consuming several large capsules a day. The study represents the first attempt to determine if betaine, an alternative compound within the same metabolic pathway but with a much lower molecular weight, also increases serum choline levels. As the first step, this proposal seeks to address this in non-pregnant women. Specifically, the goals are to (a) assess whether changes in serum choline levels in response to molar equivalent supplementation of phosphatidylcholine versus betaine are similar, and (b) whether, for betaine, there is a dose response relationship between supplementation dose and serum choline levels.

ELIGIBILITY:
Inclusion Criteria:

1. premenopausal
2. No nicotine use
3. No marijuana use
4. No illicit substance use
5. Weight >= 90 pounds

Exclusion Criteria:

1. self-reported body odor of unknown etiology
2. personal or family history of cystathionine beta synthase deficiency (homocystinuria)
3. personal or family history of trimethylaminuria, renal or liver disease, Parkinson's disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
change in serum choline | 4 hours post supplement.- baseline

SECONDARY OUTCOMES:
change in serum choline | 2 hours post supplementation.- baseline
change in serum choline | 6 hours post supplementation.- baseline
change in serum choline | 8 hours post supplementation.- baseline
change in serum choline | 10 hours post supplementation.- baseline
change in serum choline | 12 hours post supplementation - baseline
change in serum choline | 1 week post supplementation - baseline

CONTACTS AND LOCATIONS:
Overall Officials: Camille Hoffman, MD, Principal Investigator — Denver Health and Hospitals; Randal G Ross, MD, Study Director — University of Colorado School of Medicine; Ann Olincy, MD, Study Director — University of Colorado School of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States